CLINICAL TRIAL: NCT06567691
Title: Endoscopic Gastroenterostomy Versus Surgical Gastrojejunostomy for Treatment of Malignant Gastric Outlet Obstruction: a Randomized Controlled Trial
Brief Title: Endoscopic Gastroenterostomy Versus Surgical Gastrojejunostomy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Patrick Yachimski, Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 240747
Record Dates: First submitted 2024-08-20; First posted 2024-08-23 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Malignant Gastric Outlet Obstruction

STUDY DESIGN:
Masking Description: Due to the nature and means of access of the two interventions (one via peroral approach and one via abdominal incision) blinding of the subjects, study investigators, and treating clinicians will not be practicable short of subjecting patients to sham endoscopy and/or surgery, which we feel would be unethical.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EUS Gastrojejunostomy (Active Comparator): Patient will undergo an Endoscopic Ultrasound (EUS) Gastrojejunostomy procedure
  Interventions: Procedure: EUS Gastrojejunostomy; Other: Gastric Outlet Obstruction Scoring System (GOOSS)
- Surgical Gastrojejunostomy (Active Comparator): Patient will undergo Surgical Gastrojejunostomy procedure.
  Interventions: Procedure: Surgical Gastrojejunostomy; Other: Gastric Outlet Obstruction Scoring System (GOOSS)

INTERVENTIONS:
Procedure: EUS Gastrojejunostomy — Endoscopic Ultrasound (EUS) Gastrojejunostomy. Under live real-time EUS visualization, a solution of normal saline or water and dilute methylene blue will be infused through the nasobiliary drainage catheter to mechanically distend the small intestine and create a suitable, expanded fluid-filled target for transgastric access. Once a suitable target has been identified, a lumen apposing metal stent (LAMS) will then be deployed securely across the newly created gastroenterostomy tract. Appropriate stent placement will be confirmed.
  Arms: EUS Gastrojejunostomy
Procedure: Surgical Gastrojejunostomy — Gastrojejunostomy will be performed via an open technique using an upper midline or left sub-costal incision (at the discretion of the surgeon). An antecolic, pro-peristaltic, gastrojejunostomy will be performed using one of two standard techniques: 1) hand-sewn: 2-layer anastomosis using absorbable suture or 2) stapled: single-layer anastomosis using a surgical stapler with closed staple height ranging from 1.0 - 1.5 mm and suture closure of the common enterotomy. Feeding tube placement will be at the discretion of the operating surgeon and if performed, will be performed via a Stamm technique. Abdominal fascial closure will be performed with absorbable, monofilament, suture and skin will be closed using staples or suture at the discretion of the surgeon.
  Arms: Surgical Gastrojejunostomy
Other: Gastric Outlet Obstruction Scoring System (GOOSS) — A previously validated instrument for assessing tolerance of oral intake.

SUMMARY:
Recent comparative data suggest that EUS gastroenterostomy offers more durable patency than enteral stents for treatment of malignant GOO, leading some endoscopists to suggest that EUS gastroenterostomy should be the preferred endoscopic treatment approach.

EUS gastroenterostomy and surgical gastrojejunostomy have been compared in retrospective cohort analysis, suggesting a high technical success rate a shorter hospital length of stay for the endoscopic approach [4]. Comparison of these techniques has not been reported in controlled prospective fashion. A prospective trial is necessary in order to define the optimal interventional management option for treatment of malignant GOO in the context of the contemporary and rapidly evolved range of available endoscopic and surgical treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Able to provide informed consent
* Biopsy-proven cancer
* Cancer without surgical resection as a curative treatment option
* Clinical and radiographic presentation consistent with primary or metastatic tumor causing foregut obstruction at the level of the pylorus and/or duodenum

Exclusion Criteria:

* Age <18 years
* Pregnancy
* Unable to provide informed consent
* White Blood Count < 3,000
* Absolute Neutrophil Count < 1,500
* International normalized ratio > 1.6
* Platelet count < 100,000
* Cancer with surgical resection as a curative treatment option
* Surgically altered foregut anatomy
* Multifocal intestinal obstruction
* Abdominal ascites prohibitive of surgical candidacy
* Abdominal wall mesh prohibitive of surgical candidacy
* Child's Class B or C cirrhosis
* Gastroesophageal varices or known portal hypertension
* Body mass index >40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Compare of restoration of oral intake following EUS versus surgical gastrojejunostomy | 1 day post-operative
  A GOOSS score of 0 will be defined as intolerant of oral intake, while any GOOSS score greater than 0 will be defined as tolerant of oral intake.
  0: no oral intake
  1. oral liquids only
  2. soft solids
  3. low residue or full diet This will be given to subjects
Compare post procedure length of hospital stay | 14 days post-operative
  This outcome will be measured as the length of hospital stay (in days) from study intervention to discharge. Any accrued hospital stay from admission prior to study intervention will not be included in this assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Yachimski, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No